CLINICAL TRIAL: NCT01637402
Title: A Phase II Study of Increased-Dose Abiraterone Acetate in Patients With Castration Resistant Prostate Cancer (CRPC)
Brief Title: A Phase II Study of Increased-Dose Abiraterone Acetate in Patients With Castration Resistant Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Terence Friedlander, MD (Other)
Collaborators: Janssen Biotech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Terence Friedlander, MD, Assistant Clinical Professor, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 12551; NCI-2012-02079 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2012-07-06; First posted 2012-07-11 (Estimated); Results first posted 2020-08-17 (Actual); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: Castration Resistant Prostate Cancer
Keywords: CRPC; Prostate; Cancer
MeSH Terms: conditions — Neoplasms | interventions — Abiraterone Acetate; Prednisone

STUDY DESIGN:
Intervention Model Description: Simon's 2 stage minimax design for accrual.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standard Dose (Experimental): 1000 milligrams (mg) abiraterone acetate in combination with prednisone taken once a day until progression defined by RECIST criteria OR by the Prostate Cancer Working Group 2 (PCWG) criteria
  Interventions: Drug: Abiraterone Acetate; Drug: Prednisone
- Escalated Dose (Experimental): Participants who progressed on the standard dose will be assigned 1000 milligrams (mg) abiraterone acetate in combination with prednisone taken twice a day for at least 12 weeks until progression as defined by RECIST criteria OR by the Prostate Cancer Working Group 2 (PCWG) criteria
  Interventions: Drug: Abiraterone Acetate; Drug: Prednisone

INTERVENTIONS:
Drug: Abiraterone Acetate — Standard dose participants:
  1,000 mg, once daily, oral administration.
  Dose escalation participants:
  1,000 mg, twice daily, oral administration
  Other Names: Zytiga
Drug: Prednisone — 5 mg, twice daily, oral administration

SUMMARY:
The purpose of this study is to find out what effects, good and/or bad,an increased dose of Abiraterone Acetate in combination with prednisone has on patients and their prostate cancer. This study will investigate whether an increased-dose (2,000mg daily) is safe and potentially effective when given to patients whose cancer has grown while taking the standard dose.

DETAILED DESCRIPTION:
This is a phase II multicenter trial of Abiraterone Acetate (AA) in patients with progressive prostate cancer despite androgen deprivation with a particular focus on the pharmacokinetic, pharmacodynamic, and pharmacogenomic events occurring at the time of apparent drug resistance. All eligible patients will have baseline (prior to taking the first dose of Abiraterone Acetate 1000mg/daily) measures of routine clinical variables along with measurements of baseline and treatment related changes in testosterone, androgen, and endocrine levels, genotyping of single-nucleotide polymorphisms (SNP) in the selected enzymes known to be directly inhibited by Abiraterone Acetate, and collection of circulating tumor cells. All patients will be requested to consent for biopsies which will be performed prior to treatment and at the time of disease progression on standard dose Abiraterone Acetate therapy. These biopsies will be analyzed for expression of an androgen receptor (AR)-signature as well as for microarray analysis to explore changes in methylation, and expression of CYP17A1 and other androgen synthesis genes.

Subjects will then begin daily oral therapy with Abiraterone Acetate 1000mg po daily with physiologic prednisone 5mg BID replacement. No food should be consumed for at least 2 hours before the dose of Abiraterone Acetate and for at least 1 hour after the dose of Abiraterone Acetate is taken. Prostate-specific antigen (PSA) will be followed monthly. Abiraterone Acetate will be supplied by Janssen Services. At the end of the first month, the third month, and then every three months thereafter, Abiraterone Acetate, testosterone, and androgen levels will be followed. Subjects not achieving a greater than or equal to 30% PSA decline at 12 weeks will be taken off study. At the time of progression (defined by RECIST criteria OR by the Prostate Cancer Working Group 2 (PCWG) criteria as a 25% increase in PSA above the nadir and an increase in the absolute value PSA of at least 2ng/dl or back to baseline confirmed at least 2 weeks afterward) for subjects who achieved an initial greater than or equal to 30% PSA decline (referred to as Progressive Disease (PD) #1), subjects will begin taking Abiraterone Acetate 1000 mg po BID. Patients will continue to take prednisone 5mg twice a day (BID) and will continue this therapy until a second progression at which point they will be withdrawn from the study. While 1000 mg po BID is not the FDA recommended dose, it is the dose to be investigated in this study.

ELIGIBILITY:
Inclusion Criteria:

* Have signed an informed consent document indicating that the subjects understands the purpose of and procedures required for the study and are willing to participate in the study
* Be willing/able to adhere to the prohibitions and restrictions specified in this protocol
* Written Authorization for Use and Release of Health and Research Study Information has been obtained
* Male aged 18 years and above
* Able to swallow the study drug whole as a tablet
* Willing to take abiraterone acetate on an empty stomach; no food should be consumed at least two hours before and for at least one hour after the dose of abiraterone acetate is taken
* Patients who have partners of childbearing potential must be willing to use a method of birth control with adequate barrier protection as determined to be acceptable by the principal investigator and sponsor during the study and for 1 week after last study drug administration.
* Have a baseline serum potassium of ≥ 3.5 milliequivalents per litre (mEq/L)
* Have aspartate aminotransferase (AST), alanine aminotransferase (ALT), and bilirubin levels < 1.5 x upper limit of normal (ULN)
* Have a serum albumin of ≥ 3.0 g/dL
* Total bilirubin ≤ 1.5 x ULN (In patients with known Gilbert Syndrome, a total bilirubin ≤ 3.0 x ULN, with direct bilirubin ≤ 1.5 x ULN is acceptable)
* Have a platelet count of ≥ 100,000/μL
* Have an absolute neutrophil count of > 1500 cell/mm3
* Have a calculated creatinine clearance ≥ 60 mL/min
* Have a hemoglobin of ≥ 9.0 g/dL
* Have histologically confirmed adenocarcinoma of the prostate.
* No prior therapy with chemotherapy for metastatic prostate cancer.
* Have metastatic disease based on a positive bone scan or objective imaging on CT scan.
* Have ongoing gonadal androgen deprivation therapy with Luteinizing hormone-releasing hormone (LHRH) analogues or orchiectomy. Patients who have not had an orchiectomy must be maintained on effective LHRH analogue therapy for the duration of the trial.
* Testosterone < 50 ng/dL.
* Progressive disease after androgen deprivation: PSA evidence for progressive prostate cancer consists of a PSA level of at least 2 ng/ml which has risen on at least 2 successive occasions, at least 2 weeks apart. If the confirmatory PSA value is less than the screening PSA value, then an additional test for rising PSA will be required to document progression.
* Antiandrogen Withdrawal (AAWD): Patients who are receiving an antiandrogen as part of primary androgen ablation must demonstrate disease progression following discontinuation of antiandrogen.
* Disease progression after antiandrogen withdrawal is defined as 2 consecutive rising PSA values, obtained at least 2 weeks apart, or documented osseous or soft tissue progression.
* For patients receiving flutamide, at least one of the PSA values must be obtained 4 weeks or more after flutamide discontinuation.
* For patients receiving bicalutamide or nilutamide, at least one of the PSA values must be obtained 6 weeks or more after antiandrogen discontinuation.
* No antiandrogen withdrawal response is expected in patients in whom antiandrogen therapy did NOT result in a decline in PSA or in those patients in whom the response to antiandrogens was < 3 months. Therefore, it is not necessary to wait for AAWD in patients without PSA decline on an anti-androgen or in those in whom a PSA response lasted < 3 months.
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1
* Life expectancy of ≥ 12 weeks.

Exclusion Criteria:

* Active infection or other medical condition that would make prednisone/prednisolone (corticosteroid) use contraindicated
* Known brain metastasis
* Uncontrolled hypertension (systolic BP ≥ 160 mmHg or diastolic BP ≥ 95 mmHg) Patients with a history of hypertension are allowed provided blood pressure is controlled by anti-hypertensive treatment
* Active or symptomatic viral hepatitis or chronic liver disease
* History of pituitary or adrenal dysfunction
* Clinically significant heart disease as evidenced by myocardial infarction, or arterial thrombotic events in the past 6 months, severe or unstable angina, or New York Heart Association (NYHA) Class II-IV heart disease or cardiac ejection fraction measurement of < 50 % at baseline
* Atrial Fibrillation, or other cardiac arrhythmia requiring medical therapy
* Administration of an investigational therapeutic within 30 days of screening
* Have poorly controlled diabetes
* Have a history of gastrointestinal disorders (medical disorders or extensive surgery) that may interfere with the absorption of the study agents
* Have a pre-existing condition that warrants long-term corticosteroid use in excess of study dose
* Have known allergies, hypersensitivity, or intolerance to abiraterone acetate or prednisone or their excipients
* Any condition which, in the opinion of the investigator, would preclude participation in this trial.
* Pure small cell carcinoma of the prostate or any mixed histology cancer of the prostate (eg: neuroendocrine) which contains < 50% adenocarcinoma.
* Therapy with other hormonal therapy, including any dose of megestrol acetate (Megace), finasteride (Proscar), dutasteride (Avodart) any herbal product known to decrease PSA levels (e.g., Saw Palmetto and PC-SPES), or any systemic corticosteroid within 4 weeks prior to first dose of study drug.
* Prior therapy with Abiraterone Acetate or other CYP17 inhibitor(s) including TAK-700 or TOK-001, or investigational agent(s) targeting the androgen receptor for metastatic prostate cancer.
* Prior therapy with ketoconazole for > 2 weeks for prostate cancer.
* Therapy with supplements or complementary medicines/botanicals within 4 weeks of first dose of study drug, except for any combination of the following:
* Conventional multivitamin supplements
* Selenium
* Lycopene
* Soy supplements
* Prior radiation therapy completed < 4 weeks prior to enrollment
* Prior chemotherapy for castration resistant prostate cancer. Patients who have received chemotherapy for early stage prostate cancer (e.g. as part of a neoadjuvant or adjuvant trial) or for other malignancies are eligible provided that >1 year has passed since the administration of the last chemotherapy dose.
* Any "currently active" second malignancy, other than non-melanoma skin cancer. Patients are not considered to have a "currently active" malignancy, if they have completed therapy and are considered by their physician to be at least less than 30% risk of relapse over next year.
* Active psychiatric illnesses/social situations that would limit compliance with protocol requirements.
* Patients in whom urgent chemotherapy, in the opinion of the treating physician, is indicated should not be enrolled in this study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2013-03-13 (Actual); Primary Completion 2017-02-27 (Actual); Study Completion 2017-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Terence Friedlander, MD, Study Chair — University of California, San Francisco
Locations (2):
- United States (2):
  - University of California, San Francisco, San Francisco, California
  - Oregon Health and Science University, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Friedlander TW, Graff JN, Zejnullahu K, Anantharaman A, Zhang L, Paz R, Premasekharan G, Russell C, Huang Y, Kim W, Aggarwal RR, Lin AM, Fong L, Alumkal JJ, Beer TM, Sharifi N, Alyamani M, Dittamore R, Small EJ, Paris PL, Ryan CJ. High-Dose Abiraterone Acetate in Men With Castration Resistant Prostate Cancer. Clin Genitourin Cancer. 2017 Dec;15(6):733-741.e1. doi: 10.1016/j.clgc.2017.05.026. Epub 2017 Jun 3. PMID 28655452

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through the Urologic Oncology Program at University of California, San Francisco
Pre-assignment Details: All participants were prescribed the standard dose(STD). Participants who did not exhibit prostate-specific antigen (PSA) decline at 12 weeks were deemed 'primary-resistant' and taken off study. Participants continued STD until progression, at which time, they were assigned to the escalated dose was for a minimum of 12 weeks.
Groups:
- Standard Dose: Abiraterone 1000 mg once daily Prednisone 5 mg twice daily
- Escalated Dose: Abiraterone 1000 mg twice daily Prednisone 5 mg twice daily
Period: Standard Dose Regimen
Arm/Group | Standard Dose | Escalated Dose
Started | 41 | 0 (Escalated dose not introduced as treatment option until after Week 12 evaluation)
Completed | 38 | 0
Not Completed | 3 | 0
Not completed — Lack of Efficacy | 2 | 0
Not completed — Adverse Event | 1 | 0
Period: Week 12 Evaluation
Arm/Group | Standard Dose | Escalated Dose
Started | 38 | 0 (Escalated dose not introduced as treatment option until after Week 12 evaluation)
Completed | 32 | 0
Not Completed | 6 | 0
Not completed — Lack of Efficacy | 6 | 0
Period: Treatment Regiments Post Week 12
Arm/Group | Standard Dose | Escalated Dose
Started | 14 (Patients continuing on standard dose) | 18 (Patients who progressed after decline on standard dose)
Completed | 5 | 14
Not Completed | 9 | 4
Not completed — Not evaluable for response after 12wks | 0 | 4
Not completed — Withdrawal by Subject | 4 | 0
Not completed — Progression after escalation arm closed | 5 | 0

BASELINE CHARACTERISTICS:
Population: This is a sequential treatment design. Participants enrolled in standard dose continued on regimen based on disease status at week 12 evaluation and progression status. At progression, an escalated dose option was assigned based on response to standard dose. 18 of the 41 total were assigned to escalated dose regimen.
Groups:
- All Patients Who Received Treatment: Abiraterone Acetate: Standard dose: 1,000 mg, once daily, oral administration
  Increased dose offered after week 12 evaluation to participants who progressed after decline on standard dose: 1,000 mg, twice daily, oral administration
  Prednisone: 5 mg, twice daily, oral administration
Arm/Group | All Patients Who Received Treatment
Number analyzed (Participants) | 41
Age, Continuous [Median (Full Range); unit: years] | 68 [55 to 79]
Age, Continuous [Mean (Full Range); unit: years] — Population: Measure Description: This measure presents data for the 18 participants that were subsequently randomized to the second treatment arm
  years
    number analyzed (Participants) | 18
    (all) | 67.4 [55 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 37
  Unknown or Not Reported | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: This measure presents data for the 18 participants that were subsequently randomized to the second treatment arm
  Participants
    number analyzed (Participants) | 18
    Hispanic or Latino | 0
    Not Hispanic or Latino | 17
    Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 30
  More than one race | 0
  Unknown or Not Reported | 8
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: This measure presents data for the 18 participants that were subsequently randomized to the second treatment arm
  Participants
    number analyzed (Participants) | 18
    American Indian or Alaska Native | 0
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 0
    White | 16
    More than one race | 0
    Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 41
Prior Therapies [Count of Participants; unit: Participants]
  Radical Prostatectomy | 12
  Definitive Radiotherapy | 15
  Metastatic at Diagnosis | 14
Prostate Specific Antigen levels [Median (Full Range); unit: ng/dl] | 23.18 [0.4 to 1763.9]

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With PSA Response From Dose Escalation
Description: A PSA response for the dose escalation group is defined as a participant with a documented PSA decline after 12 weeks of therapy with standard-dose, then had disease progression, and then achieved a ≥30% PSA decline after 12 weeks from the start of dose escalation therapy.
Time Frame: Up to 12 weeks from start of dose escalation
Measure: Count of Participants; unit: Participants
Groups:
- Dose Escalation: Dose Escalation (until PSA decrease of at least 30% after 12 weeks):
  Abiraterone 1,000 mg, twice daily, Prednisone 5 mg twice daily
Arm/Group | Dose Escalation
Number analyzed (Participants) | 14
Participants | 0

2. Secondary Outcome: Number of Participants With Worst-grade, Treatment-related Toxicities for Dose Escalation Group
Description: Frequency of any treatment-related toxicity with increased-dose Abiraterone Acetate by maximum observed grade will be tabulated for the study cohort. Toxicities will be graded for management according to NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 as a measure of patient safety.
Time Frame: Up to 24 months
Measure: Count of Participants; unit: Participants
Groups:
- Dose Escalation (CTCAE Grade 1): Worst grade adverse event with CTCAE Grade 1 for patients taking Abiraterone 1000 mg twice daily, Prednisone 5 mg twice daily
- Dose Escalation (CTCAE Grade 2): Worst grade adverse event with CTCAE Grade 2 for patients taking Abiraterone 1000 mg twice daily, Prednisone 5 mg twice daily
- Dose Escalation (CTCAE Grade 3): Worst grade adverse event with CTCAE Grade 3 for patients taking Abiraterone 1000 mg twice daily, Prednisone 5 mg twice daily
- Dose Escalation (CTCAE Grade 4): Worst grade adverse event with CTCAE Grade 4 for patients taking Abiraterone 1000 mg twice daily, Prednisone 5 mg twice daily
Arm/Group | Dose Escalation (CTCAE Grade 1) | Dose Escalation (CTCAE Grade 2) | Dose Escalation (CTCAE Grade 3) | Dose Escalation (CTCAE Grade 4)
Number analyzed (Participants) | 18 | 18 | 18 | 18
Participants
  Dry Mouth | 1 | 0 | 0 | 0
  Hypertension | 0 | 1 | 0 | 0
  Alanine aminotransferase increase | 0 | 0 | 1 | 0
  Irritability | 0 | 1 | 0 | 0
  Aspartate aminotransferase increased | 0 | 1 | 0 | 0
  Hypokalemia | 0 | 1 | 0 | 0
  Purpura | 1 | 0 | 0 | 0
  Fatigue | 0 | 1 | 0 | 0

3. Secondary Outcome: Time to PSA Progression for Dose Escalation Cohort
Description: Time to PSA progression as defined by RECIST criteria or by the Prostate Cancer Working Group 2 (PCWG) criteria for patients whom were treated with increased dose Abiraterone Acetate.
Time Frame: up to 24 months
Measure: Median (Full Range); unit: months
Groups:
- Dose Escalation: Abiraterone 1,000 mg, twice daily, Prednisone 5 mg twice daily
Arm/Group | Dose Escalation
Number analyzed (Participants) | 14
months | 12 [6 to 14.5]

4. Secondary Outcome: Progression Free Survival for Dose Escalation Cohort
Description: Progression free survival for patients treated with increased dose Abiraterone Acetate
Time Frame: up to 24 months
Population: Progression-free survival could not be calculated due to the lack of objective response in the dose escalation group (i.e. no patients were progression-free).
Arm/Group | Dose Escalation
Number analyzed (Participants) | 0

5. Secondary Outcome: Serum Concentration Levels of Abiraterone Acetate Over Time
Description: Pharmacokinetic assessment at the initiation of standard dose therapy, at the time of initial disease progression, at the time of a response to increased dose of abiraterone acetate and at the time of disease progression on increased-dose therapy.
Time Frame: Up to 24 months
Population: Only 26 patients on the standard dose had pharmacokinetic samples available for analysis at time of first blood draw. No patients displayed a response to increased-dose therapy therefore data for concentration at time of response to increased dose was not collected.
Measure: Median (Full Range); unit: nanograms per millilitre (ng/mL)
Groups:
- Concentration at First Draw on Standard Dose Therapy (4 Weeks): Plasma Abiraterone concentration at 4 weeks for patients on standard dose
- Concentration at Time of Disease Progression on Standard Dose: Plasma Abiraterone concentration at time of disease progression on standard dose
- Concentration at Time of Response to Increased-dose: Plasma Abiraterone concentration at the time of a response to increased-dose Abiraterone Acetate
- Concentration at Time of Disease Progression on Increased Dose: Plasma Abiraterone concentration at the time of disease progression on increased-dose therapy.
Arm/Group | Concentration at First Draw on Standard Dose Therapy (4 Weeks) | Concentration at Time of Disease Progression on Standard Dose | Concentration at Time of Response to Increased-dose | Concentration at Time of Disease Progression on Increased Dose
Number analyzed (Participants) | 26 | 26 | 0 | 14
nanograms per millilitre (ng/mL) | 5.5 [1.26 to 56.2] | 14.2 [0.8 to 221] |  | 31.5 [5.2 to 148]

6. Secondary Outcome: Correlation of Circulating Testosterone Levels at Baseline and Week 12
Description: Pearson's correlation coefficients ("r") will be calculated to summarize the relationship between testosterone values at baseline and at 12 weeks. Testosterone labs will be obtained at an earlier time point if the patient comes off study for disease progression before week 12. Coefficients are on a continuous scale ranging from -1 to +1 with a value of -1 indicating a perfect negative linear association of testosterone levels between the 2 time points, a value of 0 indicating no association between testosterone levels between the two time points, and a value of +1 indicating a positive linear association of testosterone levels between the two time points.
Time Frame: Baseline and Week 12
Population: Testosterone levels were maximally suppressed below the laboratory limit of detection (LOD) at week 12 for patients on standard-dose therapy so no correlation could be performed. There were no responders in dose escalation so evaluation of hormonal changes with dose-escalated group was not pursued.
Groups:
- Standard Dose: Standard Dose until progression:
  Abiraterone 1,000 mg, once daily, Prednisone 5 mg twice daily
Arm/Group | Standard Dose | Dose Escalation
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Comparison of Circulating Testosterone Levels Between Primary-Resistant Patients and Responders
Description: The distribution of the baseline testosterone levels and the change in hormone level at 12 weeks will be compared between patients experiencing a PSA decline >30% (responders) and patients without such a PSA decline (primary-resistant) using a two group t statistic. Measurements will be obtained at an earlier time point if the patient comes off study for disease progression before week 12.
Time Frame: Baseline and Week 12
Population: Testosterone levels were maximally suppressed below the laboratory limit of detection (LOD) at week 12 for patients on standard-dose therapy so no correlation could be performed. There were no responders in the dose escalation group so evaluation of hormonal changes with dose-escalated group was not pursued.
Measure: Mean (Standard Deviation); unit: Nanograms per decilitre (ng/dL)
Groups:
- Testosterone in Primary Resistant (STD): Testosterone levels in patients without > 30% PSA decline during standard dose therapy.
- Testosterone in Responders (STD): Testosterone levels in patients with > 30% PSA decline during standard dose therapy
Arm/Group | Testosterone in Primary Resistant (STD) | Testosterone in Responders (STD)
Number analyzed (Participants) | 7 | 19
Nanograms per decilitre (ng/dL) | NA (NA) — below the level of detection | NA (NA) — below the level of detection

8. Secondary Outcome: Correlation of Circulating Dehydroepiandrosterone (DHEA) Levels From Baseline to Week 12
Description: Pearson's correlation coefficients ("r") will be calculated to summarize the relationship between DHEA values at baseline and at 12 weeks. DHEA labs will be obtained at an earlier time point if the patient comes off study for disease progression before week 12. Coefficients are on a continuous scale ranging from -1 to +1 with a value of -1 indicating a perfect negative linear association of DHEA levels between the 2 time points, a value of 0 indicating no association between DHEA levels between the two time points, and a value of +1 indicating a positive linear association of DHEA levels between the two time points.
Time Frame: Baseline and Week 12
Population: No DHEA values were collected for week 12 in dose escalation group so correlation of for dose escalation could not be performed.
Measure: Number; unit: correlation coefficient (r)
Arm/Group | Standard Dose | Dose Escalation
Number analyzed (Participants) | 26 | 0
correlation coefficient (r) | 0 |

9. Secondary Outcome: Comparison of Circulating DHEA Levels Between Primary-Resistant and Responders
Description: The distribution of the baseline DHEA levels and the change in hormone level at 12 weeks will be compared between patients experiencing a PSA decline >30% (responders) and patients without such a PSA decline (primary-resistant) using a two group t statistic. Measurements will be obtained at an earlier time point if the patient comes off study for disease progression before week 12.
Time Frame: Baseline and Week 12
Population: Twenty-six patients had both baseline and follow-up samples available for analysis. There were no responders in dose escalation group so evaluation of hormonal changes with dose-escalated group was not pursued.
Measure: Mean (Full Range); unit: ng/dL
Groups:
- DHEA in Primary Resistant (STD): DHEA levels in patients without > 30% PSA decline during standard dose therapy.
- DHEA in Responders (STD): DHEA levels in patients with > 30% PSA decline during standard dose therapy.
Arm/Group | DHEA in Primary Resistant (STD) | DHEA in Responders (STD)
Number analyzed (Participants) | 7 | 19
ng/dL
  Initial draw | 56.2 [11.2 to 223.9] | 79.4 [11.2 to 281.83]
  Progression / Week 12 | 28.5 [14.1 to 141.2] | 13.5 [3.1 to 44.7]

10. Secondary Outcome: Correlation of Circulating Dehydroepiandrosterone-sulfate (DHEA-S) Levels at Baseline and Week 12
Description: Pearson's correlation coefficients ("r") will be calculated to summarize the relationship between DHEA-S values at baseline and at 12 weeks. DHEA-S labs will be obtained at an earlier time point if the patient comes off study for disease progression before week 12. Coefficients are on a continuous scale ranging from -1 to +1 with a value of -1 indicating a perfect negative linear association of DHEA-S levels between the 2 time points, a value of 0 indicating no association between DHEA-S levels between the two time points, and a value of +1 indicating a positive linear association of DHEA-S levels between the two time points.
Time Frame: Baseline and Week 12
Population: DHEA-S levels were maximally suppressed below the laboratory limit of detection (LOD) at week 12 for patients on standard-dose therapy so no correlation could be performed. There were no responders in dose escalation so evaluation of hormonal changes with dose-escalated group was not pursued.
Groups:
- Dose-Escalation: Dose Escalation (until PSA decrease of at least 30% after 12 weeks):
  Abiraterone 1,000 mg, twice daily, Prednisone 5 mg twice daily
Arm/Group | Standard Dose | Dose-Escalation
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Comparison of Circulating DHEA-S Levels Between Primary-Resistant Patients and Responders
Description: The distribution of the baseline DHEA-S levels and the change in hormone level at 12 weeks will be compared between patients experiencing a PSA decline >30% (responders) and patients without such a PSA decline (primary-resistant) using a two group t statistic. Measurements will be obtained at an earlier time point if the patient comes off study for disease progression before week 12.
Time Frame: Baseline and Week 12
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: microgram per deciliter (µg/dL)
Groups:
- DHEA-S in Primary Resistant (STD): DHEA-S levels in patients without > 30% PSA decline during standard dose therapy.
- DHEA-S in Responders (STD): DHEA-S levels in patients with > 30% PSA decline during standard dose therapy.
Arm/Group | DHEA-S in Primary Resistant (STD) | DHEA-S in Responders (STD)
Number analyzed (Participants) | 7 | 19
microgram per deciliter (µg/dL) | NA (NA) — below the level of detection | NA (NA) — below the level of detection

12. Secondary Outcome: Correlation of Circulating Androstenedione Levels at Baseline and Week 12
Description: Pearson's correlation coefficients ("r") will be calculated to summarize the relationship between androstenedione values at baseline and at 12 weeks. Androstenedione labs will be obtained at an earlier time point if the patient comes off study for disease progression before week 12. Coefficients are on a continuous scale ranging from -1 to +1 with a value of -1 indicating a perfect negative linear association of androstenedione levels between the 2 time points, a value of 0 indicating no association between androstenedione levels between the two time points, and a value of +1 indicating a positive linear association of androstenedione levels between the two time points.
Time Frame: Baseline and Week 12
Population: Androstenedione levels were maximally suppressed below the laboratory limit of detection (LOD) at week 12 for patients on standard-dose therapy so no correlation could be performed. There were no responders in dose escalation so evaluation of hormonal changes with dose-escalated group was not pursued.
Arm/Group | Standard Dose | Dose Escalation
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Comparison of Circulating Androstenedione Levels Between Primary-Resistant Patients and Responders
Description: The distribution of the baseline androstenedione levels and the change in hormone level at 12 weeks will be compared between patients experiencing a PSA decline >30% (responders) and patients without such a PSA decline (primary-resistant) using a two group t statistic. Measurements will be obtained at an earlier time point if the patient comes off study for disease progression before week 12.
Time Frame: Baseline and Week 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: ng/dL
Groups:
- Androstenedione in Primary Resistant (STD): Androstenedione levels in patients without > 30% PSA decline during standard dose therapy.
- Androstenedione in Responders (STD): Androstenedione levels in patients with > 30% PSA decline during standard dose therapy.
Arm/Group | Androstenedione in Primary Resistant (STD) | Androstenedione in Responders (STD)
Number analyzed (Participants) | 7 | 19
ng/dL | NA (NA) — below the level of detection | NA (NA) — below the level of detection

ADVERSE EVENTS:
Time Frame: Up to 24 months
Groups:
- Standard Dose Therapy: Abiraterone 1000 mg daily, Prednisone 5 mg twice daily
Arm/Group | Standard Dose Therapy | Dose Escalation
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/18
Serious Adverse Events (participants affected / at risk) | 7/41 | 1/18
Other Adverse Events (participants affected / at risk) | 34/41 | 10/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Dose Therapy (N=41) | Dose Escalation (N=18)
Atrial fibrillation (Cardiac disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Dental caries (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 0 | 1
Lung infection (Infections and infestations) | 0 | 1
Upper respiratory infection (Infections and infestations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Dose Therapy (N=41) | Dose Escalation (N=18)
Hypertension (Vascular disorders) | 5 | 2
Hot flashes (Vascular disorders) | 5 | 0
Vascular disorders - Other, specify (Vascular disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 4 | 0
Nausea (Gastrointestinal disorders) | 3 | 1
Dyspepsia (Gastrointestinal disorders) | 3 | 0
Vomiting (Gastrointestinal disorders) | 3 | 0
Oral pain (Gastrointestinal disorders) | 1 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 5 | 2
Pain (General disorders) | 4 | 1
Edema limbs (General disorders) | 3 | 0
Irritability (General disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 6 | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 4 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Upper respiratory infection (Infections and infestations) | 5 | 0
Skin infection (Infections and infestations) | 1 | 1
Dizziness (Nervous system disorders) | 3 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 1
Bruising (Injury, poisoning and procedural complications) | 4 | 0
Fall (Injury, poisoning and procedural complications) | 4 | 0
Fracture (Injury, poisoning and procedural complications) | 4 | 0
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 4 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Purpura (Skin and subcutaneous tissue disorders) | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 3 | 1
Cystitis noninfective (Renal and urinary disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Cataract (Eye disorders) | 0 | 1
Creatinine increased (Investigations) | 5 | 1
Alanine aminotransferase increased (Investigations) | 3 | 1
Aspartate aminotransferase increased (Investigations) | 3 | 1
Anxiety (Psychiatric disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Additional accrual to the dose-increased arm was halted early due to lack of efficacy at interim analysis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-02-17): https://cdn.clinicaltrials.gov/large-docs/02/NCT01637402/Prot_SAP_000.pdf